CLINICAL TRIAL: NCT01042626
Title: Dissimilar PTH, Gastrin, and Ionized Calcium Response to Oral Peptones in Normocalcemic Primary Hyperparathyroidism, Hypercalcemic Primary Hyperparathyroidism and Healthy Subjects
Brief Title: Oral Peptones Load in Normocalcemic and Hypercalcemic Primary Hyperparathyroidism and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Piedmont (Other)
Collaborators: University of Milan (Other)
Responsible Party: Maurizio Bevilacqua, L. Sacco Hospital (Vialba)
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NO012010
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Hyperparathyroidism; Hypercalcemia
Keywords: Receptors, Calcium sensing; Parathyroid Hormone
MeSH Terms: conditions — Hyperparathyroidism; Hypercalcemia

ARMS (3):
- Normocalcemic Hyperparathyroidism (Experimental)
  Interventions: Other: Oral peptones load
- Hypercalcemic Hyperparathyroidism (Experimental)
  Interventions: Other: Oral peptones load
- Healthy subjects (Active Comparator)
  Interventions: Other: Oral peptones load

INTERVENTIONS:
Other: Oral peptones load — Enrolled subjects will receive 10 g Liebig meat extract diluted in 250ml of 0.9% saline

SUMMARY:
The purpose of this study is to assess if subjects with hyperparathyroidism with normal serum calcium levels have different responses in the calcium regulating hormonal handling compared to a) patients with primary hyperparathyroidism and high serum calcium levels; b) healthy subjects.

The differences will be evaluated with oral peptones load and subsequent blood samples collected every 15 minutes for two hours. Ionized calcium, phosphate, gastrin and PTH levels will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. normocalcemic hyperparathyroidism

   * presence of high serum levels of intact PTH
   * serum ionized calcium levels in the high normality range
2. hypercalcemic hyperparathyroidism

   * presence of high serum levels of intact PTH
   * high serum ionized calcium levels

Exclusion Criteria:

1. potential causes of secondary hyperparathyroidism like renal insufficiency, liver disease, malabsorption, hypercalciuria, Paget's disease, thiazide diuretic or lithium use.
2. bone disease of any origin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
PTH levels variations | 2 hours
Ionized serum calcium variations | 2 hours
Serum phosphate variations | 2 hours
Serum gastrin variations | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- L. Sacco Hospital (Vialba), Milan, MI, Italy

REFERENCES:
- [Background] Bevilacqua M, Dominguez LJ, Righini V, Valdes V, Vago T, Leopaldi E, Baldi G, Barrella M, Barbagallo M. Dissimilar PTH, gastrin, and calcitonin responses to oral calcium and peptones in hypocalciuric hypercalcemia, primary hyperparathyroidism, and normal subjects: a useful tool for differential diagnosis. J Bone Miner Res. 2006 Mar;21(3):406-12. doi: 10.1359/JBMR.051210. Epub 2005 Dec 19. PMID 16491288